CLINICAL TRIAL: NCT02707705
Title: Premedication With an Auricular Acupuncture Protocol in Elective Cesarean Section .
Brief Title: Preoperative Auricular Acupuncture in Elective Cesarean Section.
Acronym: CESAUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 69HCL15_0352
Record Dates: First submitted 2016-02-23; First posted 2016-03-14 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Reduction, Elective Cesarean Section
MeSH Terms: interventions — Disinfection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- : Auricular Acupuncture (needle patch) group A (Experimental): Needle patch: Patients receiving the auricular acupuncture protocol with needles inserted on adhesive tape.
  Interventions: Device: Apply an auricular acupuncture protocol by stimulating specific points of the ear with needles inserted on adhesive tape (Pyonex®).; Procedure: Disinfection
- Needle-free patch: group P. (Placebo Comparator): Patients who received the auricular acupuncture protocol with adhesive tape without needles.
  Interventions: Device: Apply a device having no real effect; Procedure: Disinfection
- No intervention: group C (No Intervention): Patients without any device or intervention.

INTERVENTIONS:
Device: Apply an auricular acupuncture protocol by stimulating specific points of the ear with needles inserted on adhesive tape (Pyonex®). — Intervention Description :
  The auricular acupuncture protocol is based on an anxiolytic triad of three points selected according to the World Health Organization classification. These points are detected and located precisely by a differential detector starting with the right ear, and in the absence of response, the points are searched on the left ear. The detected points are treated by application of adhesive tape with needles of diameter 0.2 mm and length 0.9 mm.
  Data collected :
  * T0 : anxiety VAS, pain VAS, APAIS, ANI, arterial pressure and cardiac frequency
  * T1 : anxiety VAS, pain VAS, APAIS, ANI, arterial pressure, cardiac frequency and side effects
  * T2 : anxiety VAS, pain VAS, arterial pressure, cardiac frequency and side effects
  * T3 : anxiety VAS, pain VAS, arterial pressure, cardiac frequency and side effects
  Arms: : Auricular Acupuncture (needle patch) group A
Device: Apply a device having no real effect — The three points of the protocol are detected and located precisely by a differential detector starting with the right ear, and in the absence of response, the points are searched on the left ear.The detected points are treated by application of adhesive tape without needle.
  Data collected :
  * T0 : anxiety VAS, pain VAS, APAIS, ANI, arterial pressure and cardiac frequency
  * T1 : anxiety VAS, pain VAS, APAIS, ANI, arterial pressure, cardiac frequency and side effects
  * T2 : anxiety VAS, pain VAS, arterial pressure, cardiac frequency and side effects
  * T3 : anxiety VAS, pain VAS, arterial pressure, cardiac frequency and side effects
  Arms: Needle-free patch: group P.
Procedure: Disinfection — The ear is disinfected by applying Chlorhexidine®.
  Arms: : Auricular Acupuncture (needle patch) group A; Needle-free patch: group P.

SUMMARY:
Preoperative anxiety before cesarean section is common and may be severe. Stress consequences are often deleterious for the mother and for the upcoming newborn. Means to reduce anxiety before cesarean section are limited. Anxiolytic drugs are avoided in the context of the birth of a newborn. Auricular acupuncture has been shown to relieve anxiety disorders. The aim of this study is to evaluate the anxiolytic effect of auricular acupuncture administered before an elective cesarean section. Anxiety will be measured at T0: inclusion (approximately 1-2 hours before cesarean section) and T1: departure to surgical unit (approximately 30 minutes to 1 hour after T0). Patches (needle or needle-free) will be set up at T0 just after the initial anxiety assessment (anxiety Visual Analog Scale aVAS).

ELIGIBILITY:
Inclusion Criteria:

* All patients American Society of Anaesthesiologists 1or 2 targeted for elective cesarean section under spinal anesthesia
* Aged over 18 years
* Affiliation to social security
* Participation Consent signed after oral and written information

Exclusion Criteria:

* Guardianship
* Psychological disorders preventing informed consent
* Long-term antidepressant or anxiolytic
* Previous history of auricular acupuncture
* Refusal of participation in the study
* Cesarean section for placenta accreta
* Presence of a pacemaker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Comparison of anxiety variation between group A (Auricular acupuncture, needle patch) and group P (needle-free patch) via visual analog scale. | measured at the inclusion (T0) and 30min/1h after inclusion (T1).
  Degree of reduction in anxiety VAS score between T0 and T1 and comparison between group A and group P. Anxiety will be assessed using a Visual Analogue Scale scoring between 0 (complete absence of anxiety) and 100 (greatest possible level of anxiety).

SECONDARY OUTCOMES:
Potential placebo effect of auricular acupuncture by measuring Anxiety variation between the 3 groups. | measured at the inclusion (T0), 30min/1h after inclusion (T1), 1h/2h after inclusion (incision T2) and 3h/4h after inclusion (back in post-operative surveillance room T3).
  Variation of anxiety VAS between T0 and T1 between the 3 groups (needle patch, needle-free patch and no intervention.
  Comparing the percentage of patients relieved by auricular acupuncture between the 3 groups (decrease of anxiety VAS score of at least 20%).
To evaluate anxiolytic effect of auricular acupuncture on anxiety measured by Amsterdam Preoperative Anxiety and Information Scale (APAIS). | measured at the inclusion (T0) and 30min/1h after inclusion (T1).
  Variation of APAIS between T0 and T1, comparison between the 3 groups. APAIS is a self-reported questionnaire comprising six questions.
To evaluate the effect of auricular acupuncture on parasympathetic tone measured by Analgesia Nociception Index (ANI). | measured at the inclusion (T0) and 30min/1h after inclusion (T1).
  Variation of ANI between T0 and T1, comparison between the 3 groups. ANI is a 0 to 100 index derived from heart rate variability which provides a continuous measurement of the parasympathetic tone.
Study of the correlation between ANI and anxiety VAS. | measured at the inclusion (T0) and 30min/1h after inclusion (T1).
  Variation of ANI between T0 and T1, comparison between the 3 groups, and correlation with anxiety VAS. ANI is a 0 to 100 index derived from heart rate variability which provides a continuous measurement of the parasympathetic tone.
To evaluate the effect of auricular acupuncture on perioperative pain. | Measured at1h/2h after inclusion (incision T2) and 3h/4h after inclusion (back in post-operative surveillance room T3).
  VAS for pain is a self-reported measure varying from, 0 (no pain) to 100 (greatest possible level of pain). A comparison of VAS score will be made between the 3 groups.
Report of potential adverse events of auricular acupuncture. | Measured at 30min/1h after inclusion (T1), 1h/2h after inclusion (incision T2) and 3h/4h after inclusion (back in post-operative surveillance room T3).
  collection of potential side effects.
Correlation between APAIS and anxiety VAS. | Measured at the inclusion (T0) and 30min/1h after inclusion (T1).
  Variation of APAIS between T0 and T1, comparison between the 3 groups, and correlation with anxiety VAS. APAIS is a self-reported questionnaire comprising six questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Favre-Felix J, Laurent V, Branche P, Huissoud C, Raffin M, Pradat P, Aubrun F, Dziadzko M. Auricular Acupuncture for Preoperative Anxiety in Parturient Women with Scheduled Cesarean Section: A Randomized Placebo-Controlled Blind Study. J Integr Complement Med. 2022 Jul;28(7):569-578. doi: 10.1089/jicm.2021.0346. Epub 2022 Apr 8. PMID 35394895